CLINICAL TRIAL: NCT00380263
Title: Basic Scientific Research Investigating PACAP38 Headache Inducing Effects in Migraine Patients
Brief Title: PACAP38´s (Pituitary Adenylate Cyclase-Activating Polypeptide) Headache Inducing Characteristics and Effects on the Cerebral Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Henrik Schytz/MD, Danish Headache Center
Other Study IDs: KA-20060087
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Last update posted 2008-05-30 (Estimated); Status verified 2008-05

CONDITIONS: Migraine Without Aura
MeSH Terms: conditions — Migraine without Aura | interventions — Pituitary Adenylate Cyclase-Activating Polypeptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: PACAP38 — 10 pmol/kg/min given one time

SUMMARY:
To investigate headache score and accompanying symptoms during and after infusion of PACAP38 i migraine patients

DETAILED DESCRIPTION:
To investigate headache score and accompanying symptoms during and after infusion of PACAP38

Changes in regional cerebral blood flow (rCBF) in the area supplied by middle cerebral artery (MCA), blood flow in MCA, diameter of the superficial temporal artery (STA) and radial artery (RA)

ELIGIBILITY:
Inclusion Criteria:

* Healthy migraine patient without aura
* Aged 18-50
* 50-100 kg
* Fertile women must use safe contraceptives (IUD, oral contraceptives, surgical sterilisation and long lasting gestagen.

Exclusion Criteria:

* Tension type headache more than five times/month
* Other primary headaches
* Daily medication except contraceptives
* Drug taken within 4 times the halflife for the specific drug except contraceptives
* Pregnant or lactating women
* Exposure to radiation within the last year
* Headache within the last 48 hours before start of trial
* Hypertension
* Hypotension
* Respiratory or cardiac disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2006-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Schytz, MD, Principal Investigator — Danish Headache Center
Locations (1):
- Dansih Headache Center, Glostrup Municipality, Denmark